CLINICAL TRIAL: NCT00980876
Title: Multicentric, Double Blind, Randomized, Parallel Comparative Study Between Ciprofloxacin HCl 2 mg/mL + Hydrocortisone 10 mg/mL Ear Suspension and Cipro HC®, for the Assessment of Efficacy and Safety in Patients With Otitis Externa.
Brief Title: A Comparative Study Between Two Formulations of the Ciprofloxacin Hydrochloride + Hydrocortisone Otic Suspension
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Farmoquimica S.A. (Industry)
Collaborators: Pharmagenix Projetos em Medicina Farmacêutica Ltda. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: STPh 09/08
Record Dates: First submitted 2009-09-18; First posted 2009-09-21 (Estimated); Last update posted 2015-04-17 (Estimated); Status verified 2012-03

CONDITIONS: Otitis Externa
MeSH Terms: conditions — Otitis Externa | interventions — ciprofloxacin, hydrocortisone drug combination; Ciprofloxacin; Hydrocortisone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cipro HC (Active Comparator): Reference product
  Interventions: Drug: Cipro HC
- Ciprofloxacin HCl and Hydrocortisone (Experimental): Test product
  Interventions: Drug: Ciprofloxacin HCl and Hydrocortisone

INTERVENTIONS:
Drug: Cipro HC — Cipro HC (Ciprofloxacin HCl and Hydrocortisone)
  Arms: Cipro HC
Drug: Ciprofloxacin HCl and Hydrocortisone — Ciprofloxacin Hydrochloride and Hydrocortisone
  Other Names: Otociriax
  Arms: Ciprofloxacin HCl and Hydrocortisone

SUMMARY:
The objective of this study is to compare the efficacy and safety profiles of the test product containing 2 mg/mL ciprofloxacin hydrochloride associated with 10 mg/mL of hydrocortisone with the reference product Cipro HC®, in patients with acute otitis externa.

DETAILED DESCRIPTION:
Phase III, non inferiority, multicentric, controlled, single blind, parallel-group, randomized study.

Population: 224 patients with external otitis , men and women aged between 1 - 70 years.

Primary endpoint: The primary endpoint of this study is the elimination of pain, swelling and otorrhea (cure).

Secondary endpoint: The endpoint will be the identification of the side effects of medication use.

ELIGIBILITY:
Inclusion Criteria:

* Informed of the nature of the study and given written informed consent;
* Patients with acute otitis externa;
* Intact tympanic membrane.

Exclusion Criteria:

* Known allergy or sensitivity to Ciprofloxacin Hydrochloride and Hydrocortisone;
* Patient has the tympanic membrane not intact;
* Diabetes
* Bilateral Acute Otitis Externa;
* Pregnant or lactating patients;
* Overt fungal Acute Otitis Externa;
* Other diseases of the ear
* Current Infection requiring systemic antimicrobial therapy.
* Current enrollment in an investigational drug or device study or participation in such a study within 30 days of entry into this study.

Ages: 1 Year to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 224 (Actual)
Dates: Start 2012-04; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Cure (reduced pain, swelling and otorrhea) | 7 days

SECONDARY OUTCOMES:
Identification of possible side effects | 7 days

CONTACTS AND LOCATIONS:
Overall Officials: Agricio N. Crespo, Phd, Principal Investigator — Clínica Quiron
Locations (1):
- Clínica Quiron, Campinas, São Paulo, Brazil